CLINICAL TRIAL: NCT04555187
Title: Cardiovascular Risk Stratification in Covid-19
Acronym: CaVaR-Co19
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Larisa Tereshchenko, Associate Professor of Medicine, Oregon Health and Science University
Other Study IDs: STUDY00021368
Record Dates: First submitted 2020-09-16; First posted 2020-09-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Cardiovascular Risk Factor
Keywords: Covid19; cardiovascular risk factor; electrocardiogram; risk stratification
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid19-positive: Covid19 test positive. age >= 18 y.
- Covid19-negative: Covid19 test negative. age >=18y

SUMMARY:
This retrospective double-cohort study seeks to:

1. Describe the cardiovascular manifestations and electrophysiological (EP) substrate in COVID-19 infection and their association with clinical outcomes; and
2. Develop a method of cardiovascular risk stratification in COVID-19

ELIGIBILITY:
Inclusion Criteria:

* age >=18y
* available data on Covid19 test in the electronic medical record (either positive or negative)

Exclusion Criteria:

* no data of Covid19 test

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records of patients who had Covid19 test performed
Sampling Method: Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Number and rate of persons with cardiovascular composite outcome | 6 months after Covid19 test
  Number and rate of persons with composite of all-cause death, critical care utilization (ICU bed), development of a life-threatening arrhythmia (ventricular tachycardia/ventricular fibrillation or sudden cardiac arrest), acute heart failure, myocardial infarction (STEMI, NSTEMI, or silent MI), or incident stroke, whichever comes first.

SECONDARY OUTCOMES:
Rate of all-cause death outcome | 6 months after covid19 test
  Rate of all-cause death outcome
Rate of cardiac arrhythmia | 6 months after covid19 test
  Rate of any documented cardiac arrhythmia (tachy - or brady- arrhythmia)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Tereshchenko, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tereshchenko LG, Bishop A, Fisher-Campbell N, Levene J, Morris CC, Patel H, Beeson E, Blank JA, Bradner JN, Coblens M, Corpron JW, Davison JM, Denny K, Earp MS, Florea S, Freeman H, Fuson O, Guillot FH, Haq KT, Kim M, Kolseth C, Krol O, Lin L, Litwin L, Malik A, Mitchell E, Mohapatra A, Mullen C, Nix CD, Oyeyemi A, Rutlen C, Tam AE, Van Buren I, Wallace J, Khan A. Risk of Cardiovascular Events After COVID-19. Am J Cardiol. 2022 Sep 15;179:102-109. doi: 10.1016/j.amjcard.2022.06.023. Epub 2022 Jul 15. PMID 35843735
- [Derived] Tereshchenko LG, Pourbemany J, Haq KT, Patel H, Hyde J, Quadri S, Ibrahim H, Tongpoon A, Pourbemany R, Khan A. An electrophysiological substrate of COVID-19. J Electrocardiol. 2023 Jul-Aug;79:61-65. doi: 10.1016/j.jelectrocard.2023.03.010. Epub 2023 Mar 20. PMID 36963283